CLINICAL TRIAL: NCT04235985
Title: Evaluation of Chlorhexidine Gluconate Concentration on Skin of Human Subjects Following
Brief Title: Evaluation of Chlorhexidine Gluconate Concentration on Skin of Human Subjects Following Multiple Application Times
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: #1906236-150B
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: General Skin Cleansing
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Intervention Model Description: Volunteer forearms will be marked with 6 test sites which will be randomly assigned a time point for the application.
Masking Description: This is a cross-over design study where it will only be possible to mask the Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All time points (Other)
  Interventions: Combination Product: Chlorhexidine Gluconate with HUBS

INTERVENTIONS:
Combination Product: Chlorhexidine Gluconate with HUBS — 4% CHG soap will be applied to HUBS following manufacturers recommendation and applied to skin for different application times as dictated by the randomization of the marked sites on the forearm. Followed by a HUBS moistened with water.

SUMMARY:
This study will evaluate the amount of chlorhexidine gluconate (CHG) present on treated skin of human volunteers following different application times with a test material bathing system. The amount of recovered CHG that resides on the skin following each of the evaluated application times will be evaluated via high performance liquid chromatography with ultraviolet detection (HPLC-UV) and correlated with the MIC values determined separately.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age and can be of either sex and of any race.
* Subjects must be able to read and understand English.
* Subjects must possess both forearms and have a minimum forearm length (wrist crease to elbow crease) of 8.25 inches [21 cm].
* Subjects must be in good general health (i.e., no current or recent severe illness) and have no medical diagnosis of mitral valve prolapse with heart murmur, congenital heart disease, an organ transplant, medicated or uncontrolled diabetes, hepatitis B or C, an immunocompromised condition such as AIDS (or HIV positive), lupus, fibromyalgia, ulcerative colitis, Crohn's disease, moderate to severe asthma (requiring daily use of medication), or medicated multiple sclerosis.

Exclusion Criteria:

* Participation in a clinical study within 7 days of participating in this study or current participation in another clinical study.
* Presence of tattoos, active skin rashes, dermatoses, or breaks in the skin of the forearms or hands. Subjects must also have no inflammatory skin conditions (such as atopic dermatitis / eczema, contact dermatitis, or psoriasis) anywhere on the body.
* Known allergies or sensitivities to latex (natural rubber), alcohols, sunscreens, deodorants, laundry detergents, inks, metals, topically-applied fragrances (e.g., colognes or perfumes), cleansers, soaps, lotions, or to common antibacterial agents particularly chlorhexidine gluconate (CHG).
* Have experienced hives (raised welts) as a reaction to anything that contacted the skin, with the exception of plants known to cause reactions for most humans (e.g., poison oak or poison ivy).
* Have a history of anaphylactic shock, anaphylactoid reaction, or anaphylactoid shock.
* Any prosthetic device or joint (e.g., pins, screws, plates, or rods) installed in the arms within the last 6 months.
* Any type of indwelling port or Peripherally-Inserted Central Catheter (PICC).
* Subject is pregnant, plans to become pregnant or impregnate a sexual partner within the pre-test and test periods of the study, or is nursing a child.
* Any medical condition or use of any medications that, in the opinion of the Principal Investigator or Consulting Physicians, should preclude participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Chlorhexidine skin levels | range from 15 to 120 seconds
  To find out how much CHG is left on the skin with different application times

CONTACTS AND LOCATIONS:
Overall Officials: Russell Griggs, Principal Investigator — BSLI
Locations (1):
- Bioscience Laboratories, Inc, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No